CLINICAL TRIAL: NCT05317520
Title: The Effect of Cold Vapor Application on Sore Throat in The Patients Extubated After Surgery: A Randomized Control Trial
Brief Title: The Effect of Cold Vapor Application on Postoperative Sore Throat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Hatice Özsoy, Lecturer, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Mehmet Akif Ersoy University
Record Dates: First submitted 2021-07-27; First posted 2022-04-07 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Sore Throat
Keywords: Extubation; Sore throat; Cold vapor; Nursing
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Intervention Model Description: Patients were divided into intervention and control groups using a simple randomized control method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Cold vapor was applied 3 times in total at 0th,2nd and 6th hours.
  Interventions: Procedure: Cold vapor
- Control group (No Intervention): No cold vapor was applied at 0th,2nd and 6th hours.

INTERVENTIONS:
Procedure: Cold vapor — The Ramsey Sedation Scale was used to assess wakefulness after patients were extubated and arrived at the recovery unit at the 0th hour postoperatively. Sore throat, localization of pain, hoarseness, dry throat, and swallowing difficulty were evaluated in patients with a score of 2 according to this scale. Sore throat of the patients was evaluated with Numerical Rating Scale. Then, cold vapor was applied for 15 minutes with a vapor machine used as a standard in the hospital by the researcher. After the cold vapor application was finished, the patients' sore throat, localization of pain, hoarseness, swallowing difficulty and dry throat were re-evaluated with the same forms.
  Sore throat were evaluated before the application of cold vapor at the 2nd and 6th hours. Then cold vapor was applied for 15 minutes. After the cold vapor application was finished, sore throat were re-evaluated.
  At the 24th hour, cold vapor was not applied to the patients. Only sore throat were evaluated.
  Arms: Intervention group

SUMMARY:
To determine the effect of cold vapor given in the post-extubation period on sore throat.

DETAILED DESCRIPTION:
General anesthesia increases the comfort of the patient by ensuring that the patient does not feel the surgical interventions and pain during the operation. The necessity of intubation is known in patients who have undergone surgery under general anesthesia. Intubation provides benefits such as keeping the airway open, controlling the airway and breathing, reducing respiratory effort and dead space volume, preventing aspiration, and facilitating resuscitation in case of any problem.

Although surgical interventions are an important treatment option for health problems, postoperative complications such as sore throat, dry throat, hoarseness and dysphagia due to laryngeal and pharyngeal traumas caused by intubation are frequently observed especially in patients receiving general anesthesia.

Although it is seen in the literature that pharmacological, non-pharmacological and herbal methods are applied to reduce postoperative sore throat, there are not enough studies examining the effect of cold steam application on sore throat. With this research, it is expected that the cold steam given in the postoperative period will contribute to the relief of sore throat.

ELIGIBILITY:
Inclusion Criteria:

* Those who accept the research
* Elective laparoscopic cholecystectomy surgery planned
* Patients in ASA I and II class
* 18 years and over
* Mallampati classification I and II
* Operation time more than 30 minutes
* Literate
* No hearing problem
* Patients without understanding difficulties

Exclusion Criteria:

* Overweight patients (Body Mass Index ≥ 40)
* Patients with sore throat and lower respiratory tract infection
* Patients with Chronic Obstructive Pulmonary Disease (COPD)
* Patients with a history of allergies
* Patients with hearing problems
* illiterate patients
* ASA classification III and above
* Mallampati classification III and IV patients
* Patients with an operation time of less than 30 minutes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Sore throat | Within an hour after surgery
  In our study, a horizontally prepared Numerical Rating Scale was used to evaluate the severity of pain. Patients participating in the study were asked to rate the severity of their sore throat on a scale of 0 to 10. The scale begins with the absence of pain (0) and ends with excruciating pain (10).
  When the patient came to the recovery unit, the severity of sore throat was evaluated before and after the application of cold vapor at 0th hour.
Sore throat | 2nd hour after surgery
  In our study, a horizontally prepared Numeric Rating Scale was used to evaluate the severity of pain. Patients participating in the study were asked to rate the severity of sore throat between 0 and 10. The scale starts with the absence of pain (0) and ends with unbearable pain (10).
  The severity of sore throat was evaluated before and after the application of cold vapor at 2nd hour postoperatively.
Sore throat | 6th hour after surgery
  In our study, a horizontally prepared Numeric Rating Scale was used to evaluate the severity of pain. Patients participating in the study were asked to rate the severity of sore throat between 0 and 10. The scale starts with the absence of pain (0) and ends with unbearable pain (10).
  The severity of sore throat was evaluated before and after the application of cold vapor at 6th hour postoperatively.
Sore throat | 24th hour after surgery
  In our study, a horizontally prepared Numeric Rating Scale was used to evaluate the severity of pain. Patients participating in the study were asked to rate the severity of sore throat between 0 and 10. The scale starts with the absence of pain (0) and ends with unbearable pain (10).
  Cold vapor was not applied to the patients at the 24th hour.. Only sore throat were evaluated.

SECONDARY OUTCOMES:
Hoarseness | Within an hour after surgery
  To assess hoarseness, patients were asked a single question, "Do you have any hoarseness in your voice now?" Participants were asked to evaluate this question with a 4-point Likert-type rating.Rating; 0 = no hoarseness, 1 = slow, hoarse voice, 2 = moderate hoarseness (clear during the interview), 3 = hoarseness (completely silent, no speech).
  When the patient came to the recovery unit, the severity of hoarseness was evaluated before and after the application of cold vapor at the 0th hour.
Hoarseness | 2nd hour after surgery
  To assess hoarseness, patients were asked a single question, "Do you have any hoarseness in your voice now?" Participants were asked to evaluate this question with a 4-point Likert-type rating. Rating; 0 = no hoarseness, 1 = slow, hoarse voice, 2 = moderate hoarseness (clear during the interview), 3 = hoarseness (completely silent, no speech).
  The severity of hoarseness was evaluated before and after the application of cold vapor at the 2nd hour postoperatively.
Hoarseness | 6th hour after surgery
  To assess hoarseness, patients were asked a single question, "Do you have any hoarseness in your voice now?" Participants were asked to evaluate this question with a 4-point Likert-type rating. Rating; 0 = no hoarseness, 1 = slow, hoarse voice, 2 = moderate hoarseness (clear during the interview), 3 = hoarseness (completely silent, no speech).
  The severity of hoarseness was evaluated before and after the application of cold vapor at the 6th hour postoperatively.
Hoarseness | 24th hour after surgery
  To assess hoarseness, patients were asked a single question, "Do you have any hoarseness in your voice now?" Participants were asked to evaluate this question with a 4-point Likert-type rating. Rating; 0 = no hoarseness, 1 = slow, hoarse voice, 2 = moderate hoarseness (clear during the interview), 3 = hoarseness (completely silent, no speech).
  Cold vapor was not applied to the patients at the 24th hour. Only hoarseness was evaluated.
Dry throat and swallowing difficulty | Within an hour after surgery
  The patients were asked to rate the severity of dry throat and swallowing difficulty between 0 and 4 (0=None, 1=Mild, 2=Moderate, 3=Extreme, 4=Unbearable).
  When the patient came to the recovery unit, the severity of throat dryness and swallowing difficulty was evaluated before and after the application of cold vapor at the 0th hour.
Dry throat and swallowing difficulty | 2nd hour after surgery
  The patients were asked to rate the severity of dry throat and swallowing difficulty between 0 and 4 (0=None, 1=Mild, 2=Moderate, 3=Extreme, 4=Unbearable).
  At the 2nd hour postoperatively, the severity of throat dryness and swallowing difficulty were evaluated before and after the application of cold vapor.
Dry throat and swallowing difficulty | 6th hour after surgery
  The patients were asked to rate the severity of dry throat and swallowing difficulty between 0 and 4 (0=None, 1=Mild, 2=Moderate, 3=Extreme, 4=Unbearable).
  At the 6th hour postoperatively, the severity of throat dryness and swallowing difficulty were evaluated before and after the application of cold vapor.
Dry throat and swallowing difficulty | 24th hour after surgery
  The patients were asked to rate the severity of dry throat and swallowing difficulty between 0 and 4 (0=None, 1=Mild, 2=Moderate, 3=Extreme, 4=Unbearable).
  Cold vapor was not applied to the patients at the 24th hour. Only dry throat and swallowing difficulty were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Özsoy, Principal Investigator — Burdur Mehmet Akif Ersoy University
Locations (1):
- Hatice Özsoy, Merkez, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: Relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.